CLINICAL TRIAL: NCT01737203
Title: Phase 1, Open-Label, Randomized, Single-Dose, 3-Way Crossover Study Assessing Bioequivalence Of Sildenafil 50 Mg Orally-Disintegrating Tablet With Or Without Water To Viagra® 50 Mg Oral Tablet With Water Under Fasted Condition
Brief Title: Bioequivalence Study For Orally-Disintegrating Tablet Of Sildenafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1481315
Record Dates: First submitted 2012-08-31; First posted 2012-11-29 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Viagra; ODT; bioquivalence
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Viagra (Active Comparator): Oral tablet of sildenafil citrate (Japanese commercial tablet: Viagra® tablet) 50 mg as a single oral dose under fasted conditions
  Interventions: Drug: Viagra
- ODT without water (Experimental): Sildenafil ODT 50 mg without water as a single oral dose under fasted conditions
  Interventions: Drug: sildenafil ODT
- ODT with water (Experimental): Sildenafil ODT 50 mg with water as a single oral dose under fasted conditions
  Interventions: Drug: sildenafil ODT

INTERVENTIONS:
Drug: Viagra — 50 mg tablet on Day 1 of each period
  Other Names: sildenafil citrate
  Arms: Viagra
Drug: sildenafil ODT — 50 mg tablet on Day 1 of each period
  Arms: ODT without water
Drug: sildenafil ODT — 50 mg tablet on Day 1 of each period
  Arms: ODT with water

SUMMARY:
The purpose of this study is to assess the bioequivalence of Sildenafil ODT 50 mg without water to Japanese commercial oral tablet of sildenafil citrate (Viagra® tablet) 50 mg under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male subjects between the ages of 20 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Baseline orthostatic hypotension defined as a >=20 mm Hg reduction in systolic blood pressure (SBP), a >=10 mm Hg reduction in diastolic blood pressure (DBP) or the development of significant postural symptoms (dizziness, lightheadedness, vertigo) when going from the supine to standing position.
* Subjects who are currently prescribed or taking nitrates or nitric oxide donors in any form on either a regular or intermittent basis.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose
Maximum Observed Plasma Concentration (Cmax) | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose
Maximum Observed Plasma Concentration (Cmax) | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose
Plasma Decay Half-Life (t1/2) | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 9 days
Diastolic and Systolic Blood Pressure | 9 days
12-lead electrocardiogram (ECG) | 9 days
Pulse rate (PR) | 9 days
Number of Participants With Laboratory Test Values of Potential Clinical Importance | 9 days
Mean Residence Time(MRT) | 0, 0.05, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481315&StudyName=Bioequivalence%20Study%20For%20Orally-Disintegrating%20Tablet%20Of%20Sildenafil